CLINICAL TRIAL: NCT04635735
Title: A Phase I/II Trial of Ipilimumab After CD34-Selected Allogeneic Stem Cell Transplantation for Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Study of Ipilimumab After Stem Cell Transplantation in People With Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-329
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Results first posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-02

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: Ipilimumab; Stem Cell Transplantation; 20-329
MeSH Terms: conditions — Multiple Myeloma | interventions — Ipilimumab

STUDY DESIGN:
Intervention Model Description: This is a phase I/II, single arm, open label trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ipilimumab After Stem Cell Transplantation (Experimental): The patient will be admitted to a single room on the Adult Transplantation Service and allogeneic CD34-selected PBSC or marrow transplantation performed as per MSKCC adult BMT guidelines. Patients will be evaluated at approximately day 100 (±2 weeks) after allo-HSCT.
  Interventions: Drug: Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab 3 mg/kg every 3 weeks for 4 doses.

SUMMARY:
This study will test the safety of ipilimumab to see what effects, if any, the drug has when used as maintenance therapy for people with relapsed/refractory multiple myeloma who have received chemotherapy and allogeneic hematopoietic stem cell transplant (AHCT). The investigators also want to find out whether giving ipilimumab after chemotherapy and AHCT is a better way to control the multiple myeloma than chemotherapy and AHCT alone.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria prior to Allogeneic Hematopoietic Stem Cell Transplantation (alloHSCT):

* Willing and able to participate as a research subject and provide informed consent (Note: an LAR may sign the consent form on the partipant's behalf)
* Diagnosis of relapsed refractory multiple myeloma defined as more than 2 lines of prior therapy with at least a very good partial remission to most recent salvage therapy.

  * Patients should have R-ISS stage II or III disease at diagnosis or high risk cytogenetics by IMWG criteria (t(4;14), del(17/17p), t(14;16), t(14;20), nonhyperdiploidy, and gain(1q)) at any time since diagnosis

Note:. A line of therapy is treatment between diagnosis and progression or between two progressions

* Eligible for CD34-selected HSCT according to MSKCC adult BMT guidelines.
* Have a 10/10 matched donor
* Age ≥ 21, < 73 years.
* Karnofsky (adult) Performance Status ≥ 70%.
* Patients must have adequate organ function measured by:

  1. Cardiac: LVEF at rest must be ≥ 50%
  2. Hepatic:

     * < 3x ULN ALT
     * < 1.5 ULN total serum bilirubin, unless there is congenital benign hyperbilirubinemia.
  3. Renal: serum creatinine <1.2 mg/dl or if serum creatinine is outside the normal range, then CrCl > 40 ml/min (measured or calculated/estimated) with dose adjustment of Fludarabine for <70ml/min
  4. Pulmonary: DLCO > 50% of predicted (corrected for hemoglobin).

Inclusion Criteria prior to Ipilimumab:

* Non progressive myeloma (partial response or better) as defined by International Myeloma Working Group (IMWG) criteria
* Engraftment of all cell lines without transfusion dependence, defined as:

  * absolute neutrophil count > 1.0K/mcL x 3 consecutive days
  * platelets > 50K/mcLx 7 consecutive days without platelet transfusion
  * no platelet or RBC transfusions within the preceding 7 days
* ≥ 80% donor chimerism in the bone marrow

Exclusion Criteria:

Exclusion Criteria prior to Allogeneic Hematopoietic Stem Cell Transplantation (alloHSCT):

* Patients ineligible for therapy with ipilimumab, for example:.

  1. Active autoimmune disease or any condition requiring systemic treatment with either corticosteroids (>10 mg daily of prednisone equivalents) or other immunosuppressive medications at enrollment. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
  2. History of motor neuropathy considered to be of autoimmune origin (e.g., Guillain-Barre Syndrome, Myasthenia Gravis).
* Female patients who are pregnant or breast-feeding.
* Patients with plasma cell leukemia at the time of diagnosis.
* Patients who have undergone prior allogeneic hematopoietic stem cell transplantation.
* Patients who have had a previous malignancy that is not in remission.

Exclusion Criteria prior to Ipilimumab:

* Active infection or treatment for infection (patients on Cytomegalovirus (CMV) therapy will be considered eligible; patients with CMV viremia by PCR or disease with end-organ involvement will not be eligible)
* Active GVHD of any grade or prior grade 3-4 GVHD
* Active immune suppression, defined as:

  * active use of calcineurin inhibitors, mycophenolate mofetil, or other immunomodulators
  * steroid dosing exceeding 10 mg/d prednisone or equivalent
* Receiving immunomodulatory agents (ex. thalidomide, lenalidomide, pomalidomide)

Ages: 21 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-01-12 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gunjan Shah, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ipilimumab After Stem Cell Transplantation
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ipilimumab After Stem Cell Transplantation
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 62 [59 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose of Ipilimumab
Description: A maximum of 12 patients will be accrued and DLTs will be assessed in these patients. If any DLT is observed in more than one of the six patient cohort, a lower dose of ipilimumab will be evaluated in a new six patient cohort.
Time Frame: 1 year
Population: Data were not collected
Arm/Group | Ipilimumab After Stem Cell Transplantation
Number analyzed (Participants) | 0

2. Primary Outcome: Phase II: Progression Free Survival (PFS)
Description: criteria of the International Myeloma Working Group
Time Frame: 2 years
Population: Data were not collected
Arm/Group | Ipilimumab After Stem Cell Transplantation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to a year
Arm/Group | Ipilimumab After Stem Cell Transplantation
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/35/NCT04635735/Prot_SAP_001.pdf